CLINICAL TRIAL: NCT01663142
Title: Early Postoperative Recurrence in Crohn's Disease: Predictors of Research Targeting the Constitutional Mutation of IRGM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 09-API-02
Record Dates: First submitted 2012-08-06; First posted 2012-08-13 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2010-05

CONDITIONS: Flammatory Bowel Disease; Crohn's Disease
Keywords: Crohn's disease; gastrointestinal tract
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lesional tissue samples and healthy in cryotubes, taken from surgical specimens or biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who receive surgical resection for intestinal in CD

SUMMARY:
Crohn's disease is a disease of complex etiology, multifactorial and still poorly understood. This disease, due to its morbidity and mortality, poses a significant public health problem in France. Apart from the involvement of bacterial factors and those involving the permeability of the epithelial barrier, it is now well recognized that several factors are associated with genetic predisposition in some of these patients. Among these factors, the Nod2 mutations were first identified. Studies concerning the presence of these mutations and the severity of disease results were sometimes conflicting. Very recently, new interesting mutations in genes involved in autophagy were found with greater frequency in patients with Crohn's disease. These mutations observed in Atg16 and IRGM genes. It has been particularly shown on large patient cohorts,the IRGM polymorphism was associated with a progressive disease, with histological severity scores. One of the severity criteria of Crohn's disease is the early recurrence observed in some patients after surgical resection of the injured segment. Predictive factors for such recurrence after surgery are not known or not.

ELIGIBILITY:
Inclusion Criteria:

* Sick in whom endoscopic control six months after surgery is needed to assess the presence and severity of endoscopic recurrence in order to alter the medical management.
* Persons affiliated to the Social Security
* Persons who have signed informed consent

Exclusion Criteria:

* Patient not affiliated to social security
* Pregnant Women
* Persons participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sick to benefit from ileal, colonic or ileocolic continuity with re Cohn proved a complicated disease (stenosis or fistula) or resistant to medical treatment well led
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Search for IRGM mutations and compare the frequency of these mutations. | 6 months post surgery
  Patients who receive surgical resection for intestinal MC have, within six months after surgery gastrointestinal endoscopy for judging the endoscopic recurrence and modify treatment if necessary. This quantifies the endoscopic recurrence of i0 to i4 classified according to the Rutgeerts score (45). Patients who have a score ≥ i2 have a severe endoscopic recurrence. We will compare the prevalence of sick with a score ≥ i2 in patient groups with or without mutation in the gene IRGM. The investigators will look for the existence of a mutation in the gene IRGM, Atg16 and IL23R. The mutation in the gene IRGM being the main prognostic factor, mutations in the genes IL23R Atg16 and prognostic factors constituting secondary.

SECONDARY OUTCOMES:
To assess the prevalence of mutations IGRM in a prospective series of 200 patients operated | 6 months post surgery
  The prevalence of mutations IGRM, Atg16 and IL23 will be determined
Determine whether there are phenotypic characteristics of the disease associated with mutations of IGRM | 6 months post surgery
  The investigators will compare the frequency of postoperative recurrence in patients who have a mutation in the genes IL23 and Atg16
Determine whether there are pathological features associated with mutations of IGRM. | 6 months post surgery
  The investigators will determine if the main phenotypic characteristics of CD (age of onset, time between diagnosis and surgery, use of immunosuppressive and biologic therapies, smoking localization of the disease, etc..) Are associated with increased prevalence of mutations of IGRM, Atg16 and IL23R.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier HEBUTERNE, PU-PH, Study Director — Centre Hospitalier Universitaire de Nice
Locations (4):
- France (4):
  - CHU de Grenoble, Grenoble
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nice, Nice